CLINICAL TRIAL: NCT01262963
Title: An Open-Label Study to Characterize the Absorption, Distribution, Metabolism and Elimination of a Single Oral 14C Labeled Dose of GSK2118436 in Subjects With BRAF Mutant Solid Tumors
Brief Title: An Absorption, Distribution, Metabolism and Excretion (ADME) Study of Single Oral Dose [14C] GSK2118436 in Subjects With BRAF Mutant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113463
Record Dates: First submitted 2010-12-02; First posted 2010-12-20 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: GSK2118436; BRAF inhibitor; BRAF positive tumor; ADME; Oncology
MeSH Terms: conditions — Neoplasms | interventions — dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Medication (Experimental): GSK2118436 suspension
  Interventions: Drug: GSK2118436

INTERVENTIONS:
Drug: GSK2118436 — A single oral dose of 95 mg of GSK2118436 containing approximately 80 µCi of radioactivity

SUMMARY:
The study is a Phase 1, open-label study designed to characterize the absorption, distribution, metabolism and excretion of GSK2118436 following administration of a single oral 14C labeled dose of GSK2118436 as a suspension in subjects with BRAF mutation positive tumors.

DETAILED DESCRIPTION:
GSK2118436 is an orally administered, potent and selective small molecule BRAF inhibitor that is being developed for the treatment of BRAF mutation-positive tumors. The study is a Phase 1, open-label study designed to characterize the absorption, distribution, metabolism and excretion of GSK2118436 following administration of a single oral 14C labeled dose of GSK2118436 as a suspension in subjects with BRAF mutation positive tumors. A sufficient number of subjects will be enrolled to complete approximately four subjects. Following completion of the study, subjects may continue dosing with GSK2118436 in the rollover study, BRF114144.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age at the time of signing the informed consent form;
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form;
* Body weight >= 45 kg and a body mass index (BMI) >/= 19 kg/m2 and </= 35 kg/m2 (inclusive);
* Able to swallow and retain oral medication;
* BRAF mutation-positive tumor (V600 E/K mutation) as determined via relevant genetic testing;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 [Oken, 1982]; NOTE: Subjects with an ECOG performance status of 2 may be eligible with the approval of the GSK Medical Monitor
* Women of child-bearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control. Additionally, women of childbearing potential must have a negative serum pregnancy test within 14 days prior to the first dose of study treatment;
* Must have adequate organ function as defined by the following values:
* Absolute neutrophil count (ANC) >/=1.2 x 10^9/L
* Hemoglobin >/=9 g/dL
* Platelets >/=100 x 10^9/L
* Serum bilirubin </=1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) </= 2.5 x ULN; <5 x ULN if liver metastases are present (with approval of GSK medical monitor)
* Serum creatinine </= ULN or calculated creatinine clearance >/= 60 mL/min
* Prothrombin time (PT)/International normalized ratio (INR) and partial thromboplastin time (PTT) </=1.3 x ULN
* Left ventricular ejection fraction </= institutional lower limit of normal by ECHO

Exclusion Criteria:

* Currently receiving cancer therapy (e.g., chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, or major surgery) within the last three weeks; chemotherapy regimens without delayed toxicity within the last two weeks; or use of an investigational anti-cancer drug within four weeks preceding the first dose of GSK2118436;
* Current use of a prohibited medication or requires any of these medications during the study;
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice from seven days prior to the first dose of study medication;
* Current use of therapeutic warfarin (note: low molecular weight heparin and prophylactic low-dose warfarin are permitted);
* History of sensitivity to heparin or heparin-induced thrombocytopenia;
* The radiation exposure from the previous three year period is over 10 millisieverts (mSv) for subjects who have been exposed to ionizing radiation above background as a result of their work with radiation as Category A (classified) workers or as a result of research studies they may have been involved in. Subjects will be excluded if exposure levels cannot be verified. Clinical (therapeutic or diagnostic) exposure will not be included;
* An occupation which requires monitoring for radiation exposure, nuclear medicine procedures or excessive x-rays within the past 12 months;
* Any major surgery within the last four weeks;
* Unresolved toxicity equal to or greater than National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI CTCAE v4.0) [NCI, 2009] Grade 2 from previous anti-cancer therapy except alopecia;
* Presence of active gastrointestinal disease or other condition (e.g., gastrectomy, bariatric surgery, small bowel or large bowel resection) that may interfere significantly with the absorption of drugs. If clarification is needed as to whether a condition will significantly affect absorption of drugs, contact the GSK medical monitor for permission to enroll the subject;
* A history of known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with laboratory evidence HBV clearance may be enrolled with permission of the GSK medical monitor);
* Patients with a history of malignancy that have been definitively treated can be enrolled with approval of the GSK medical monitor;
* Subjects with brain metastases are excluded if their brain metastases are either:

Symptomatic Treated (surgery, radiation therapy) but not clinically and radiographically stable one month after local therapy, or Asymptomatic and untreated but > 1 cm in the longest dimension Patients with small (</= 1 cm in the longest dimension), asymptomatic brain metastases that do not need immediate local therapy can be enrolled with the approval of the GSK medical monitor. Subjects on a stable dose of corticosteroids for more than one month, or those who have been off corticosteroids for at least two weeks can be enrolled with approval of the GSK medical monitor. Subjects must also be off of enzyme-inducing anticonvulsants for more than four weeks;

* History of alcohol or drug abuse within six months prior to screening;
* Corrected QT (QTc) interval >/= 480 msecs;
* History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 24 weeks;
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; abnormal cardiac valve morphology documented by echocardiogram (subjects with minimal abnormalities [ie, mild regurgitation/stenosis] can be entered on study with approval from the GSK medical monitor); or history of known cardiac arrhythmias (except sinus arrhythmias) within the past 24 weeks;
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drugs, or excipients (note: to date there are no known drugs chemically related to GSK2118436 which are approved by the Food and Drug Administration);
* Uncontrolled medical conditions (e.g., diabetes mellitus, hypertension), psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol;
* Subjects with known glucose 6 phosphate dehydrogenase (G6PD) deficiency;
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, five half-lives or twice the duration of the biological effect of the investigational product (whichever is longer);
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period;
* Pregnant females as determined by positive pregnancy test at screening or prior to dosing;
* Lactating females who are actively breast feeding;
* Subject is mentally or legally incapacitated;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-01-26 (Actual); Primary Completion 2011-04-08 (Actual); Study Completion 2011-04-08 (Actual)

PRIMARY OUTCOMES:
• Excretion of radioactivity in urine following oral administration of [14C]GSK2118436 | Pre-dose, and post-dose for a minimum of 96 hours, and a maximum of 240 hours after dosing.
• Excretion of radioactivity in feces following oral administration of [14C]GSK2118436 | Pre-dose, and post-dose for a minimum of 96 hours, and a maximum of 240 hours after dosing.

SECONDARY OUTCOMES:
• Quantity of GSK2118436 metabolites in plasma | Pre-dose, and up to 48 hours post dose.
• Potential covalent binding of drug-related material to plasma proteins | Pre-dose, and up to 48 hours post dose.
• Blood total radioactivity | Pre-dose, and post-dose for a minimum of 96 hours, and a maximum of 240 hours after dosing.
• Blood:plasma ratio of total drug-related material (radioactivity) | Pre-dose, and post-dose for a minimum of 96 hours, and a maximum of 240 hours after dosing.
• Area under the plasma-concentration time curve (AUC) of plasma GSK2118436 and metabolites | Pre-dose, and up to 48 hours post dose.
• Number of subjects with adverse events as a measure of safety and tolerability | From date of dosing until transition to rollover protocol BRF114144 (approximately 4 - 11 days) or study follow up visit if subject does not transition to BRF114144 (approximately 14 - 21 days)
• Quantity of GSK2118436 metabolites in feces | Pre-dose, and post-dose for a minimum of 96 hours, and a maximum of 240 hours after dosing.
• Quantity of GSK2118436 metabolites in urine | Pre-dose, and post-dose for a minimum of 96 hours, and a maximum of 240 hours after dosing.
• Character of GSK2118436 metabolites in plasma | Pre-dose, and up to 48 hours post dose.
• Character of GSK2118436 metabolites in feces | Pre-dose, and post-dose for a minimum of 96 hours, and a maximum of 240 hours after dosing.
• Character of GSK2118436 metabolites in urine | Pre-dose, and post-dose for a minimum of 96 hours, and a maximum of 240 hours after dosing.
• Plasma total radioactivity | Pre-dose, and post-dose for a minimum of 96 hours, and a maximum of 240 hours after dosing.
• Maximum plasma concentration (Cmax) of plasma GSK2118436 and metabolites | Pre-dose, and up to 48 hours post dose
• Time to Cmax (Tmax) of plasma GSK2118436 and metabolites | Pre-dose, and up to 48 hours post dose
• Terminal half-life (t1/2) of plasma GSK2118436 and metabolites | Pre-dose, and up to 48 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tacoma, Washington, United States

REFERENCES:
- [Background] Bershas DA, Ouellet D, Mamaril-Fishman DB, Nebot N, Carson SW, Blackman SC, Morrison RA, Adams JL, Jurusik KE, Knecht DM, Gorycki PD, Richards-Peterson LE. Metabolism and disposition of oral dabrafenib in cancer patients: proposed participation of aryl nitrogen in carbon-carbon bond cleavage via decarboxylation following enzymatic oxidation. Drug Metab Dispos. 2013 Dec;41(12):2215-24. doi: 10.1124/dmd.113.053785. Epub 2013 Oct 4. PMID 24097902
- See also: Results for study 113463 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113463?search=study&search_terms=113463#rs